CLINICAL TRIAL: NCT00955123
Title: Effects of Prednisolone and Infliximab on the Regulation of Urea Synthesis in Patients With Active Ulcerative Colitis and Crohn's Disease
Brief Title: Effects of Prednisolone and Infliximab on the Regulation of Urea Synthesis in Active Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Karen Louise Thomsen, Dr., University of Aarhus
Other Study IDs: FHNC-KLT
Record Dates: First submitted 2009-08-03; First posted 2009-08-07 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Inflammation; Urea synthesis; Catabolism; Nitrogen balance
MeSH Terms: conditions — Inflammatory Bowel Diseases; Inflammation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma and urine.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Active inflammatory bowel disease: Patients with moderate to severe active inflammatory bowel disease (ulcerative colitis and Crohn's disease)

SUMMARY:
Loss of total mass of muscles (catabolism) is a serious clinical problem in patients with active inflammatory bowel disease (IBD). The investigators have earlier shown that the liver plays an important role in this stress-catabolism by increasing the production of urea during the inflammatory process.

The purpose of this study is to examine the effect of the anti-inflammatory drugs prednisolone and infliximab on the regulation of the urea synthesis in patients with active ulcerative colitis and Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe active inflammatory bowel disease

Exclusion Criteria:

* Viral or bacterial infections
* Other chronical inflammatory diseases
* Cancer
* Other catabolic diseases
* Treatment with prednisolone or infliximab within the last 8 weeks

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with active inflammatory bowel disease seen in the out-patients' clinic or admitted to hospital for treatment.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-01; Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Functional Hepatic Nitrogen Clearance | Before and one week after treatment

SECONDARY OUTCOMES:
Clinical and biochemical measures of inflammation | Before and one week after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Karen Louise Thomsen, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Medicine V, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Hjortebjerg R, Thomsen KL, Agnholt J, Frystyk J. The IGF system in patients with inflammatory bowel disease treated with prednisolone or infliximab: potential role of the stanniocalcin-2 / PAPP-A / IGFBP-4 axis. BMC Gastroenterol. 2019 Jun 3;19(1):83. doi: 10.1186/s12876-019-1000-6. PMID 31159802